CLINICAL TRIAL: NCT04600193
Title: a Randomized Controlled Trial of the Intake of Organic and Inorganic Phosphate in Peritoneal Dialysis Patients
Acronym: RCTOIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Stine Kristensen (Unknown); Gita Krüger Mørch (Unknown); Rizwan Butt (Unknown); Ditte Hansen (Unknown)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate professor at the university of Copenhagen, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IOOAIOP
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phosphate modified diet with organic phosphate (Experimental)
  Interventions: Other: Diet containing organic phosphate
- Phosphate modified diet with inorganic phosphate (Experimental)
  Interventions: Other: Diet containing inorganic phosphate

INTERVENTIONS:
Other: Diet containing organic phosphate — The patients will be receiving a 5 days diet containing organic phosphate
  Arms: Phosphate modified diet with organic phosphate
Other: Diet containing inorganic phosphate — The patients will be receiving a 5 days diet containing inorganic phosphate
  Arms: Phosphate modified diet with inorganic phosphate

SUMMARY:
Hyperphosphatemia is a common problem among patientens suffering from chronic kidney disease. Hyperphosphatemia is associated with increased risk of cardiovascular diseases. One of the treatments are through the diet, where patients are instructed ind reducing their daily intake of phosphate. But since phosphate exists in both organic and inorganic forms in the diet, this leads to several problems. Informations of the bioavability and furthermore the effect of plasma koncentrations of phosphate are lacking for both forms of phosphate.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Competent
* The patient should be able to take a sample of p-fluid and urine by himself
* Chronic peritoneal dialysis
* Reads and understand danish
* Has been informed written and oraly about the study and signed informed consent
* P-phosphate koncentrations 0,7-2,0 .mol/l
* P - ioniset calcium 1,1-1,4 mmol/l

Exclusion Criteria:

* Pregnant or breast-feeding
* Terminal patients
* If the experience acute infections or other acute situations they will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-03-17 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of phosphate | six days

SECONDARY OUTCOMES:
Changes in p-phosphate | six days
changes in p-calcium | six days
Changes in p-sodium | six days
Changes in p-potassium | six days
changes in p-PTH | six days
Changes in p-FGF23 | six days
Changes in p-magnesium | six days
Koncentration of phosphate in peritoneal dialysis fluid | six days
Koncentration of phosphate in urine | six days

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Herlev Hospital, Herlev, Denmark